CLINICAL TRIAL: NCT05172622
Title: A Dose-randomized, Double-blind, Placebo-controlled, Single- and Multiple-dose, Dose-escalation, Phase I Clinical Trial to Investigate the Safety, Tolerability, and Pharmacokinetic and Pharmacodynamic of JP-2266 in Healthy Subjects
Brief Title: Safety, Tolerability, and Pharmacokinetic and Pharmacodynamic Characteristics of JP-2266 in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jeil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JP-2266-101-FIH
Record Dates: First submitted 2021-11-01; First posted 2021-12-29 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JP-2266 (Experimental): Drug: JP-2266
  Interventions: Drug: JP-2266
- JP-2266 Placebo (Placebo Comparator): Drug: JP-2266 Placebo
  Interventions: Drug: JP-2266 Placebo

INTERVENTIONS:
Drug: JP-2266 — * Single Ascending Dose: Single administration on Day 1
  * Food effect cohort: Single administration on Day 1 of each period
  * Multiple Ascending Dose: Repeated administrations from D1 to D15
  Arms: JP-2266
Drug: JP-2266 Placebo — * Single Ascending Dose: Single administration on Day 1
  * Food effect cohort: Single administration on Day 1 of each period
  * Multiple Ascending Dose: Repeated administrations from D1 to D15
  Arms: JP-2266 Placebo

SUMMARY:
Phase I Clinical Trial to Investigate the Safety, Tolerability, and Pharmacokinetic and Pharmacodynamic Characteristics of JP-2266 after Oral Administration in Healthy Male Caucasian Subjects

DETAILED DESCRIPTION:
A Dose-randomized, Double-blind, Placebo-controlled, Single- and Multiple-dose, Dose-escalation, Phase I Clinical Trial to Investigate the Safety, Tolerability, and Pharmacokinetic and Pharmacodynamic Characteristics of JP-2266 after Oral Administration in Healthy Male Caucasian Subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy male Caucasian subject aged 18 to 50 years inclusive
* Body Mass Index (BMI) between 18 and 27 kg/m2 inclusive and body weight ≥ 50 kg at screening
* Signing a written informed consent prior to selection;

Exclusion Criteria:

* Any history (including family history) or presence of cardiovascular, pulmonary, gastro-intestinal, hepatic, renal, metabolic, haematological, neurologic, psychiatric, systemic or infectious disease;

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Inclusion Criteria:
  * Healthy male Caucasian subject aged 18 to 50 years inclusive
Enrollment: 80 (Estimated)
Dates: Start 2020-11-24 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
The evaluation of the number of adverse events and the number and percentage of subjects | up to Day 10
  Single Ascending Dose
Assessment of PK parameter: Maximum plasma concentration (Cmax) | up to 72hours of each period
  Food effect cohort
The evaluation of the number of adverse events and the number and percentage of subjects | up to Day 19
  Multiple Ascending Dose

CONTACTS AND LOCATIONS:
Locations (1):
- OPTIMED clinical research, Gières, France

IPD SHARING:
Plan to Share IPD: No